CLINICAL TRIAL: NCT01372878
Title: MA-204: Evaluation of Capsule Endoscopy With PillCam® COLON 2 in Visualization of the Colon
Brief Title: Evaluation of Capsule Endoscopy With PillCam® COLON 2 in Visualization of the Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: MA-204
Record Dates: First submitted 2011-06-05; First posted 2011-06-14 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2012-07

CONDITIONS: CRC Screening
Keywords: Polyps; Capsule endoscopy; Colonoscopy
MeSH Terms: conditions — Polyps | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PillCam® COLON 2 procedure — Subjects will undergo a PillCam® COLON 2 procedure which includes ingestion of the PillCam® COLON 2 capsule. PillCam® COLON 2 is a disposable, ingestible capsule that takes video images throughout the digestive system.
Procedure: Colonoscopy — Subjects will undergo standard Colonoscopy procedure 4-6 weeks after PillCam® COLON 2 procedure.
  Standard colonoscopy involves placement of a standard endoscope (a thin, flexible plastic tube) into the anus and into the colon, a tiny camera in the endoscope allows the study doctor to see the surface of the colon.

SUMMARY:
This study was design to establish the effectiveness of PillCam® Platform with the PillCam® COLON 2 capsule as demonstrated by the identification of subjects with polyps as compared to optical colonoscopy.

DETAILED DESCRIPTION:
This multi-center study was designed to evaluate the safety and effectiveness of PillCam Platform with the PillCam COLON 2 capsule as demonstrated by the identification of subjects with polyps, compared to optical colonoscopy.

884 subjects participated in this study. All subjects that were enrolled in this study were indicated and scheduled to undergo colonoscopy based on their age and demographics for screening for polyps.

Each subject was required to follow a bowel preparation regimen and to undergo capsule endoscopy (CE) followed by optical colonoscopy (OC). The optical colonoscopy procedure was scheduled 4-6 weeks after CE procedure to allow for the central readers reading of the PillCam RAPID video.

The colonoscopist was kept blinded to the CE results

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 - 75 years of age, and is classified as average risk per the AGA Guidelines on CRC Screening.
2. Subject received an explanation about the nature of the study and agrees to provide written informed consent.

Exclusion Criteria:

1. Subject has a history of colorectal cancer
2. Subjects with history of any positive colon assessment (including CT, optical colonoscopy, sigmoidoscopy etc.)
3. Subject with history of negative colon assessment (including CT, optical colonoscopy, sigmoidoscopy etc.) < 5 years as these subjects would be defined not requiring screening in this time frame
4. Subject has a first degree relative diagnosed with colorectal cancer before the age of 60 years old or 2 (or more) first degree relatives diagnosed with colorectal cancer at any age.
5. Subject is suspected or diagnosed with familial adenomatous polyposis, hereditary non polyposis colon cancer, or any high risk genetic syndrome.
6. Subject is suspected or diagnosed with inflammatory bowel disease, or chronic ulcerative colitis or Crohn's disease.
7. Subject is suspected or diagnosed with hematochezia, melena, Fe deficiency anemia or any other rectal bleeding, including positive FOBT test of any variety.
8. Subject is suspected or diagnosed with bowel obstruction.
9. Subject has dysphagia or any swallowing disorder.
10. Subject has congestive heart failure.
11. Subject has Type 1 or Type II Diabetes.
12. Subject has had prior abdominal surgery of the gastrointestinal tract in the last 6 months, other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
13. Subject has a cardiac pacemaker or other implanted electro medical device.
14. Subject has any allergy or other known contraindication to the medications used in the study.
15. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
16. Subject with any condition believed to have an increased risk for capsule retention such as intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy.
17. Subject with strictures, fistulas and/or chronic constipation.
18. Subject with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.
19. Subject with known gastrointestinal motility disorders.
20. Subject has known delayed gastric emptying.
21. Subject has any condition, which precludes compliance with study and/or device instructions.
22. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
23. Subject suffers from life threatening conditions.
24. Concurrent participation in another clinical trial using any investigational drug or device.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Prof., Principal Investigator — Indiana University Hospital, Indianapolis, IN, USA
Locations (17):
- United States (11):
  - Alabama Digestive Disorders Center P.C., Huntsville, Alabama
  - Indiana University Hospital, Indianapolis, Indiana
  - Louisville Gastroenterology Associates, Louisville, Kentucky
  - Specialists in Gastroenterology, St Louis, Missouri
  - Research Associates of New York, New York, New York
  - UNC Chapel Hill Gastroenterology and Hepatology, Chapel Hill, North Carolina
  - Dayton Gstroenterology Inc., Dayton, Ohio
  - Franklin Gastroenterology, PLLC, Franklin, Tennessee
  - Gastroenterology Consultants, P.A., Houston, Texas
  - Pasadena Gastroenterology Associates, P.A., Pasadena, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Bikur Holim Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center at Tel-Hashomer, Tel Litwinsky

REFERENCES:
- [Derived] Rex DK, Adler SN, Aisenberg J, Burch WC Jr, Carretero C, Chowers Y, Fein SA, Fern SE, Fernandez-Urien Sainz I, Fich A, Gal E, Horlander JC Sr, Isaacs KL, Kariv R, Lahat A, Leung WK, Malik PR, Morgan D, Papageorgiou N, Romeo DP, Shah SS, Waterman M. Accuracy of capsule colonoscopy in detecting colorectal polyps in a screening population. Gastroenterology. 2015 May;148(5):948-957.e2. doi: 10.1053/j.gastro.2015.01.025. Epub 2015 Jan 22. PMID 25620668

RESULTS

PARTICIPANT FLOW:
Groups:
- Colon Capsule Endoscopy, Then Standard Colonoscopy: Capsule endoscopy was ingested following colon preparation without colon insufflation or sedation.The purpose was to detect patients with polyps equal or larger than 6mm. Patients subsequently had standard colonoscopy as "gold standard" comparison
Period: Overall Study
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Started | 884
Completed | 700
Not Completed | 184
Not completed — Withdrawal by Subject | 63
Not completed — Protocol Violation | 17
Not completed — incomplete study procedure | 104

BASELINE CHARACTERISTICS:
Population: CRC population
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Number analyzed (Participants) | 884
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.29 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 487
  Male | 397
Region of Enrollment [Number; unit: participants]
  United States | 558
  Israel | 326

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of PillCam Platform With the PillCam COLON 2 Capsule in Detecting Patients With Polyps ≥6 mm Where OC Considered as the Gold Standard Reference
Description: Sensitivity and specificity of PillCam Platform with the PillCam COLON 2 capsule in detecting subjects with polyps equal to or larger than 6 mm. For a given polyp, a match between the PillCam Colon 2 Capsule and optical colonoscopy was considered if the polyp size was assessed within plus or minus 50% of the size of the estimate of the OC measurement and the polyp as appearing within the same colon segment or in adjacent segments. The polyp size measurement by optical colonoscopy was used as the reference standard.
  Sensitivity measures the proportion of actual positives which are correctly identified as such.
  Specificity measures the proportion of negatives which are correctly identified as such.
  positive event defined as patients with polyps ≥6 mm detected by OC procedure.
Time Frame: 1 year, same as study duration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Number analyzed (Participants) | 700
percentage of participants
  sensitivity of patients with Polyp>= 6 mm | 69 [63 to 74]
  specificty of patients with Polyp>= 6 mm | 87 [85 to 89]

2. Secondary Outcome: Sensitivity and Specificity of PillCam Platform With the PillCam COLON 2 Capsule in Detecting Patients With Polyps ≥10 mm Where OC Considered as the Gold Standard Reference
Description: Sensitivity and specificity of PillCam Platform with the PillCam COLON 2 capsule in detecting subjects with polyps equal to or larger than 6 mm. For a given polyp, a match between the PillCam Colon 2 Capsule and optical colonoscopy was considered if the polyp size was assessed within plus or minus 50% of the size of the estimate of the OC measurement and the polyp as appearing within the same colon segment or in adjacent segments. The polyp size measurement by optical colonoscopy was used as the reference standard.
Time Frame: 1 year, same as study duration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Number analyzed (Participants) | 700
percentage of participants
  sensitivity of patients with Polyp>= 10 mm | 64 [55 to 73]
  specificity of patients with Polyp>= 10 mm | 95 [94 to 96]

ADVERSE EVENTS:
Arm/Group | Colon Capsule Endoscopy, Then Standard Colonoscopy
Serious Adverse Events (participants affected / at risk) | 1/884
Other Adverse Events (participants affected / at risk) | 110/884
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colon Capsule Endoscopy, Then Standard Colonoscopy (N=884)
abdominal pain related to OC procedure (Gastrointestinal disorders) | 1 (1) — The event was resolved the following day
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colon Capsule Endoscopy, Then Standard Colonoscopy (N=884)
Adverse event related to preperation (Gastrointestinal disorders) | 101 (128) — adverse events were reported as related to the colon preparation such as vomiting and nausea
Adverse event related to Capsule endoscopy (Gastrointestinal disorders) | 3 (3) — Three adverse events were reported as related to the capsule procedure and resolved within the same day (i.e., severe gagging reflex, mild vomiting and abdominal cramping)
Adverse event related to Colonoscopy (Gastrointestinal disorders) | 6 (11) — Eleven adverse events were reported as related to the colonoscopy procedure such as fever, headache, abdominal pain, bloating and nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No